CLINICAL TRIAL: NCT02095236
Title: Evaluation of Inter- and Intrafractional Motion of Liver Tumors Using Interstitial Markers and Implantable Electro-magnetic Radiotransmitters in the Context of Image-guided Radiotherapy (IGRT) - the ESMERALDA Trial
Brief Title: Evaluation of Intrafractional Motion of Liver Tumors Using Markers
Acronym: ESMERALDA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative barriers
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: The ESMERALDA Trial
Record Dates: First submitted 2014-03-04; First posted 2014-03-24 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Tumor; Effects of; Movement; Radiation; Lesion
MeSH Terms: conditions — Neoplasms | interventions — Organ Motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental (Experimental): Radioopaque fiducial markers or electro-magnetic transponders will be implanted into or in close proximity of the tumor. During a radiotherapy treatment session image and/or signal acquisition will be performed by ultrasound, computed tomography, magnetic resonance imaging or by specialized signal detectors The data will help to characterize tumor and organ motion during one treatment session which may in fact have impact on dose distribution
  Interventions: Behavioral: organ motion

INTERVENTIONS:
Behavioral: organ motion — Three-dimensional intrafractional motion of a fiducial marker or a transponder during a radiotherapy treatment session. Image and/or signal acquisition will be performed by ultrasound, computed tomography, magnetic resonance imaging or by specialized signal detectors.

SUMMARY:
Radioopaque fiducial markers or electro-magnetic transponders will be implanted into or in close proximity of the tumor. During a radiotherapy treatment session image and/or signal acquisition will be performed by ultrasound, computed tomography, magnetic resonance imaging or by specialized signal detectors The data will help to characterize tumor and organ motion during one treatment session which may in fact have impact on dose distribution

DETAILED DESCRIPTION:
With the development of more conformal and precise radiation techniques such as Intensity-Modulated Radiotherapy (IMRT), Stereotactic Body Radiotherapy (SBRT) and Image-Guided Radiotherapy (IGRT), patients with hepatic tumors could be treated with high local doses by sparing normal liver tissue. However, frequently occurring large HCC tumors are still representing a dosimetric challenge in spite of modern high sophisticated RT modalities. This interventional clinical study has been set up to evaluate the value of different fiducial markers, and to use the modern imaging methods for further treatment optimization using physical and informatics approaches.Radioopaque fiducial markers or electro-magnetic transponders will be implanted into or in close proximity of the tumor. During a radiotherapy treatment session image and/or signal acquisition will be performed by ultrasound, computed tomography, magnetic resonance imaging or by specialized signal detectors The data will help to characterize tumor and organ motion during one treatment session which may in fact have impact on dose distribution

ELIGIBILITY:
Inclusion Criteria:

* indication for high precision radiotherapy of primary and secondary liver tumors using IGRT (image-guided radiotherapy)
* age ≥ 18 years of age
* ability of subject to understand character and individual consequences of the clinical trial
* written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patients to take part in the study
* medical reasons impeding marker implantation or IGRT for treatment of liver tumors.
* non-compliance of patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Three-dimensional intra- and interfractional measurement of fiducial marker or transponder motion | One treatment session for one dataset
  Three-dimensional intrafractional motion of a fiducial marker or a transponder will be recorded and analyzed during radiotherapy. Image and/or signal acquisition will be performed by ultrasound, computed tomography, magnetic resonance imaging or by specialized signal detectors. The data will help to characterize tumor and organ motion during one treatment session which may in fact have impact on dose distribution. Prediction of tumor motion is the prerequisite for innovative adaptive radiotherapy techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E Combs, MD, Principal Investigator — Department of Radiooncology, University Hospital of Heidelberg, INF 400, 69120 Heidelberg, Germany
Locations (1):
- University Hospital, Heidelberg, Germany